CLINICAL TRIAL: NCT02010528
Title: Diabetes Distress,Psychological Well-being and Family Hardiness in Parents of Children and Adolescents With Type 1 Diabetes
Brief Title: Diabetes Distress, Psychological Well-being and Family Hardiness in Parents of Children and Adolescents With T1D
Status: Completed | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: Slovenian Research Agency (ARRS) (Unknown)
Responsible Party: Principal Investigator, Tadej Battelino, Head, Dept. of Pediatric Endocrinology, Diabetes & Metabolism, University Children's Hospital, UMCL, University Medical Centre Ljubljana
Other Study IDs: DIS-PSY-PAR-T1D-2013
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-02

CONDITIONS: Type 1 Diabetes
Keywords: Diabetes related distress, children, T1D, family hardiness, psychological well-being
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Psychological Well-Being

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Type 1 diabetes: Parents or caregivers of children and adolescents with type 1 diabetes
- Controls: Parents or caregivers of children and adolescents without diabetes

SUMMARY:
Parents have an important role in child's diabetes management. Many studies show that parental psychological stress and family dynamics are associated with parental diabetes-related distress and treatment outcomes among children and adolescents with type 1 diabetes.

The aim of this study is to analyze diabetes distress (diabetes-related parenting burden and fear of hypoglycemia), parental psychological well-being (anxiety, satisfaction with life, positive and negative affect and adult attachment relationship pattern), family hardiness and characteristics of children with type 1 diabetes in a sample of mothers and fathers of children and adolescents with type 1 diabetes of ages up to 18 years.

In this study it is hypothesized that:

1. greater parental fear of hypoglycemia and diabetes-related burden are associated with lower family hardiness and worse psychological well-being parents and higher HbA1c levels in children and adolescents with type 1 diabetes;
2. mothers will report greater fear of hypoglycemia, diabetes-related burden and lower psychological well-being comparing to fathers.
3. parents of children and adolescents with type 1diabetes will report greater anxiety, lower psychological well-being and family hardiness comparing to parents of children without diabetes.

Standardized and validated questionnaires will be used to determine: parental fear of hypoglycemia, diabetes-related burden, parent level of anxiety, psychological well-being, adult attachment relationship pattern and family hardiness.

The investigators will also measure parent daily involvement in child's diabetes management, frequency of blood glucose monitoring and parent general satisfaction with glycemic control. Objective measures such as child's HbA1c level and experience of severe hypoglycemia episode will also be obtained. These measures will be correlated with other research variables.

ELIGIBILITY:
Inclusion Criteria:

* Parents or caregivers of children and adolescents with T1D of ages up to 18 years
* Minimal 1 year duration of Type 1 diabetes

Exclusion Criteria:

* Parents or caregivers of children and adolescents with T1D of ages over 18 years

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All children that have diabetes in Slovenia are controlled at the Dept. of Pediatric Endocrinology, Diabetes & Metabolism, University Children's Hospital, UMCL and the population will be taken from here
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
parental diabetes-related distress | 1 month
  To examine associations between diabetes-related distress - diabetes burden (Problem Areas In Diabetes-Parent (PAID-P) questionnaire), fear of hypoglycemia (Hypoglycemia Fear Survey-Parent (HFS-P) questionnaire, Hypoglycemia Fear Survey- Parents of Young Children (HFS-PYC) questionnaire)

SECONDARY OUTCOMES:
psychosocial characteristics | 1 month
  STAIX (State Trait Anxiety Inventory), PANAS (The Positive And Negative Affect Schedule), SWLS (Satisfaction With Life Scale), RQ (Relationship Questionnaire)

OTHER OUTCOMES:
family hardiness | 1 month
  FHI (Family Hardiness Index)
objective measures | 1 month
  * parent daily involvement in child's diabetes management
  * frequency of blood glucose monitoring
  * parent general satisfaction with glycemic control
  * child's HbA1c level
  * child's experience of severe hypoglycemia

CONTACTS AND LOCATIONS:
Overall Officials: Tadej Battelino, Study Chair — Dept. of Pediatric Endocrinology, Diabetes & Metabolism, University Children's Hospital, UMCL
Locations (1):
- Dept. of Pediatric Endocrinology, Diabetes & Metabolism, University Children's Hospital, UMCL, Ljubljana, Slovenia